CLINICAL TRIAL: NCT03039062
Title: Serum miR-122 as a Real-time Detection Biomarker of Drug-induced Liver Injury by Chemotherapy. - an Open , Multicenter, Non-interventional Clinical Trial
Brief Title: Serum miR-122 as a Real-time Detection Biomarker of Drug-induced Liver Injury by Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: LQ003
Record Dates: First submitted 2017-01-08; First posted 2017-02-01 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-01

CONDITIONS: Chemotherapeutic Toxicity; Malignant Tumor; Liver Injury
Keywords: Serum miR-122; drug-induced liver injury by chemotherapy; malignant tumor patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum miR-122 and serum ALT, AST,ALP and total bilirubin level
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Chemotherapy group: A total of 120 malignant tumor patients who need to receive chemotherapy are involved for miR-122 detection. They are from 3 centers, 40 for each center. For the first cycle of chemotherapy, the investigators will collect 0.5-1ml blood from the remained blood sample after routine blood test during chemotherapy for each patient.Each patient will have a routine blood test before(±3 days) each cycle of chemotherapy and 7(±3)days after chemotherapy. A routine blood test will include the test of ALT,AST,ALP and TBIL. Sample collection will stop after 4 cycles of chemotherapy. All blood samples collected by investigators are the remained sample after routine tests. Patients in routine care will also have blood tests before each cycle and on day 7(+/- 3) of each cycle of chemotherapy. These patients will also have blood test at these time points even if they are not in this trial.
- Healthy population: Twenty healthy women or men who come to hospitals for annual physical examinations are enrolled in this study for miR-122 detection. Investigators will collect 0.5-1 ml blood from the remained blood samples after routine blood tests during their annual physical examinations.
- Patients of intensive care unit: Fourty patients are enrolled in this group for miR-122 detection. The investigators will collect 0.5-1ml blood from the remained blood samples of their routine blood tests or when they need blood tests.

SUMMARY:
This is an open , multicenter, interventional clinical trial to conform the role of of miR-122 a real-time detection biomarker of drug-induced liver injury by chemotherapy.

DETAILED DESCRIPTION:
The endorsed standard serum biomarkers, like ALT, AST, total bilirubin, are not tissue-specific, and cannot detect drug-induced liver injury (DILI) at a very early stage, thus unable to properly guide risk assessment and patient management. miR-122 is a liver-enriched miRNA. Many studies have demonstrated that miR-122 is a sensitive and specific biomarker when DILI occurred. However, there is a lack of a standard quantification method for miR-122 and confirmatory studies using a comprehensive list of drugs and patients. The investigators have developed the miRNA-derived Fragment Length Polymorphism (miRFLP) assay for the simultaneous quantification of multiple miRNAs.The methodology improves detection reliability by eliminating intra-assay variables. In this study, the investigators will investigate the role of miR-122 as a real-time detection biomarker of drug-induced liver injury utilizing the miRFLP assay. In addition, the investigators will try to identify the normal physiological range of miR-122 in healthy population and the relationship of miR-122 and hepatic failure in patients of intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

For all the participants:

* Normal liver function biomarkers including ALT,AST,ALP,TBIL before recruitment.
* Patients with liver disease:hepatitis B，hepatitis C，cirrhosis, hepatic failure and so on.

For patients in chemotherapy group:

* Life expectancy at least 12 weeks
* 40 patients received epirubicin-containing chemotherapY
* 40 patients received paclitaxel-containing chemotherapy
* Patients received carboplatin-containing chemotherapy.
* Patients with congestive heart failure
* Unstable angina pectoris
* Previous history of myocardial infarction within 6 month prior to study entry
* Uncontrolled hypertension as determined by the Investigator or high risk uncontrolled, arrhythmia.

Exclusion Criteria:

* Patients previously received chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We recuit 3 groups of people: people with malignant tumor who will receive their first cycle of chemotherapy, healthy population and patients in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Relationship of serum miR-122 level and DILI or hepatic failure | 1 year
  Serum miR-122 level (copies/uL) and liver function (such as ALT, AST, ALP, and bilirubin levels) will be tested before and after each cycle of chemotherapy, and the relationship of serum miR-122 level fluctuation and liver injury will be investigated.

SECONDARY OUTCOMES:
Normal physiological range of miR-122 in healthy population | 1 years
  To determine a primary normal physiological range of serum miR-122 level (copies/uL) in a group of 20 healthy women and/or men.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD,PHD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, ChineseAMS, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No